CLINICAL TRIAL: NCT05583643
Title: Syringeable Atorvastatin Loaded Eugenol Enriched PEGylated Cubosomes In-situ Gel for the Intra-pocket Treatment of Periodontitis: Statistical Optimization and Clinical Assessment
Brief Title: Clinical & Biochemical Effect of Atorvastatin in Nano Particles Gel in Periodontitis Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Heba Amin Elgendy, Teaching assistant - Pharmaceutics Department - Faculty of Pharmacy, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWA00025577
Record Dates: First submitted 2022-10-13; First posted 2022-10-18 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Periodontitis
Keywords: Periodontitis; Non-surgical treatment; Atorvastatin; Phase 1 therapy
MeSH Terms: conditions — Periodontitis | interventions — Atorvastatin; Tooth Exfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 therapy (Other)
  Interventions: Other: Scaling and debridement only
- Phase 1 therapy with atorvastatin loaded into cubosomal in-situ gel (Active Comparator)
  Interventions: Drug: Atorvastatin Calcium
- Phase 1 therapy with atorvastatin loaded into in-situ gel (Active Comparator)
  Interventions: Drug: Atorvastatin Calcium

INTERVENTIONS:
Drug: Atorvastatin Calcium — Atorvastatin loaded into nano particles in-situ gel adjunctive to scaling and debridement
  Arms: Phase 1 therapy with atorvastatin loaded into cubosomal in-situ gel
Drug: Atorvastatin Calcium — Atorvastatin loaded into in-situ gel adjunctive to scaling and debridement
  Arms: Phase 1 therapy with atorvastatin loaded into in-situ gel
Other: Scaling and debridement only — Scaling and debridement only
  Arms: Phase 1 therapy

SUMMARY:
Periodontitis is a destructive chronic inflammatory disease characterized by periodontium damage and pocket formation between the tooth and the gingival margin resulting in ultimate tooth loss. Various topical anti-inflammatory drugs were used to treat inflammation in periodontitis. Introducing atorvastatin as a novel remedy for periodontitis treatment necessitates developing a syringeable modified delivery system capable of targeting inflammation within the periodontal pockets.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients
* Patients with moderate periodontitis

Exclusion Criteria:

* Pregnant women
* Lactating women
* Patients with chronic diseases

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Probing depth | 6 weeks
Bleeding index | 6 weeks
Plaque index | 6 weeks

SECONDARY OUTCOMES:
Assessment of transforming growth factor in gingival crevicular fluid | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University for Science and Technology (MUST), Giza, Egypt

IPD SHARING:
Plan to Share IPD: No